CLINICAL TRIAL: NCT02497092
Title: Effect of Different Injection Techniques on Pain Level in Intravitreal Injections
Brief Title: Different Intravitreal Injection Techniques and Pain Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Amir Sternfeld, MD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 0021-15-RMC
Record Dates: First submitted 2015-07-07; First posted 2015-07-14 (Estimated); Last update posted 2016-04-19 (Estimated); Status verified 2016-04

CONDITIONS: Injection Site Discomfort

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Slow angled injection (Active Comparator): Slow and angled insertion of the needle through the sclera
  Interventions: Other: Technique of injection
- Slow straight injection (Active Comparator): Slow and straight insertion of the needle through the sclera
  Interventions: Other: Technique of injection
- Fast angled injection (Active Comparator): fast and angled insertion of the needle through the sclera
  Interventions: Other: Technique of injection
- Fast straight injection (Active Comparator): fast and straight insertion of the needle through the sclera
  Interventions: Other: Technique of injection

INTERVENTIONS:
Other: Technique of injection

SUMMARY:
The purpose of this study is to determine whether certain intravitreal injection techniques cause less pain than others and would therefore be beneficial for the patient's well being.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving intravitreal anti vascular endothelial growth factor (VEGF) injections
* Informed consent

Exclusion Criteria:

* Dementia or any other reason for cognitive deterioration
* Technical limitations not allowing injecting by the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Pain during the injection as measured by the "Pain numeric rating scale" | Up to 2 minutes after the injection

CONTACTS AND LOCATIONS:
Overall Officials: Amir Sternfeld, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel